CLINICAL TRIAL: NCT03896048
Title: Continuous Measurement of Diaphragm Excursion as a Predictor of Extubation Failure
Status: Completed | Type: Observational
Sponsor: Respinor AS (Industry)
Collaborators: European Commission (Other)
Responsible Party: Sponsor
Other Study IDs: DM-CS-004
Record Dates: First submitted 2019-03-27; First posted 2019-03-29 (Actual); Last update posted 2021-06-14 (Actual); Status verified 2021-06

CONDITIONS: Respiration, Artificial
Keywords: diaphragm ultrasound; mechanical ventilation; diaphragm function
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Successful extubation
- Failed extubation: Failed extubation will be defined as a patient who in the first 48 hours after extubation are reintubated, have unplanned non-invasive ventilation (NIV) or who have a tracheostomy.

SUMMARY:
Background: Patients are put under invasive mechanical ventilation (MV) during respiratory failure because they can no longer breathe in a way that delivers enough oxygen to their body. MV involves placing a tube into the wind pipe that is attached to a machine (known as a ventilator) which helps the patient breathe. However, MV is associated with complications such as shrinkage and damage of the diaphragm muscle fibres. It has been shown that the diaphragm (the main breathing muscle which provides approximately 70% of the work in healthy persons) can be affected after only 3-4 days of MV. Disconnection from the ventilator (a process known as extubation) is conducted with the calculated risk that the patient may become exhausted due to the additional workload of breathing off the ventilator resulting in needing to be reconnected to the ventilator (a process known as reintubation). Reintubation requires additional deep sedation of the patient and leads to longer time connected to the ventilator, increased risk of new lung infections, prolonged stay in the intensive care unit (ICU) and further immobilisation. Thus, the intensive care physician must constantly evaluate the need for MV to maintain adequate breathing versus withdrawal as quickly as possible to reduce the risk associated with long-term use of MV. However, to date, there is no technique for continuous assessment of diaphragm function that can be easily used at the patient's bedside. RESPINOR DXT, which offers continuous ultrasound monitoring of the right diaphragm velocity without the need of the continued presence of an operator, could offer an interesting solution.

Aim: The primary objective of this study is to compare diaphragm excursion values obtained around a 30-minute SBT using RESPINOR DXT in patients who are successfully and unsuccessfully extubated. Data analysis will be performed using post-processing. The timepoints to be analysed will be:

* Pre-SBT: 10, 30 and 60 minutes before the start of the SBT
* During the 30-minute SBT: 0, 1, 2, 3, 4, 10, 20 and 30 minutes
* Post-SBT: 5, 10, 20, 30 minutes, 1, 2, 3, 4, 6, 8, 12, 24, 48 hours after the end of the 30-minute SBT.

Hypothesis: The investigators hypothesise that there will be significantly different median diaphragm excursion between successful and failed extubation groups in at least one of the timepoints of interest. The information from this pilot study will be used to design a fully-powered observational study.

Primary outcome: Median diaphragm excursion

ELIGIBILITY:
Inclusion Criteria:

* Older than 17 years,
* At least 24 hours and maximum of 7 days of invasive controlled mechanical ventilation prior to commencing pressure support ventilation,
* A minimum 30-minute SBT is planned to be initiated by the ICU physicians in charge on or before the 14th day of MV, before extubation is considered,
* The reason for admission to the ICU is adequately treated and the general condition is steadily improving, defined as reduction of general supportive ICU therapy, e.g. fluid supplements, cardiovascular stabilising medications, sedative agents, oxygen supply below 50% and mechanical ventilator support,
* Informed consent to participate in the study from patient or the close relative/next to kin.

Exclusion Criteria:

* Central or spinal neurological injury influencing central ventilation or its transmission, including critical illness neuropathy and myopathy,
* Diagnosed chronic neuromuscular disease prior to admission,
* Administration of neuromuscular blocking agents within the previous 24 hours,
* Known paralysis of a hemidiaphragm or suspicion of paralysis of a hemidiaphragm, defined by the radiographic evidence of elevation of a dome >2.5 cm compared to the contralateral dome,
* Patient with therapeutic limitation, i.e. reduced expectancy to survive,
* Women known to be pregnant,
* Protected adult who is not legally responsible and has a legal guardian,
* Skin damage or dressing at the subcostal area at the site of the probe placement.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients on mechanical ventilation in the intensive care unit for greater than 24 hours and who are considered by the treating physician to be eligible for a 30-minute spontaneous breathing trial (SBT).
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2019-03-25 (Actual); Primary Completion 2020-02-03 (Actual); Study Completion 2020-10-13 (Actual)

PRIMARY OUTCOMES:
Differences in median diaphragm excursion between patients who are successfully and unsuccessfully extubated | Up to 48 hours post-extubation

SECONDARY OUTCOMES:
Differences in maximum diaphragm excursion between patients who are successfully and unsuccessfully extubated | Up to 48 hours post-extubation
Thresholds for diaphragm excursion, rapid shallow breathing index (RSBI) and modified RSBI (m-RSBI) to predict extubation or weaning outcome at selected timepoints | Up to 48 hours post-extubation
  Thresholds for continuous diaphragm excursion, RSBI and m-RSBI will be defined by receiver operating characteristic (ROC) curve analysis to predict extubation failure. The sensitivity, specificity, positive and negative predictive value as well as the area under the ROC curves (AUROC) will be presented
Differences in median diaphragm excursion between patients who are successfully and unsuccessfully weaned | Up to 48 hours post end of SBT
  Failed weaning will be defined as a patient who fails extubation, fails the SBT or who is not extubated following a successful SBT
Differences in maximum diaphragm excursion between patients who are successfully and unsuccessfully weaned | Up to 48 hours post end of SBT

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Bergum, MD, Principal Investigator — St Olav's Hospital
Locations (1):
- St Olav's Hospital, Trondheim, Norway

REFERENCES:
- [Background] Jiang JR, Tsai TH, Jerng JS, Yu CJ, Wu HD, Yang PC. Ultrasonographic evaluation of liver/spleen movements and extubation outcome. Chest. 2004 Jul;126(1):179-85. doi: 10.1378/chest.126.1.179. PMID 15249460
- [Background] Spadaro S, Grasso S, Mauri T, Dalla Corte F, Alvisi V, Ragazzi R, Cricca V, Biondi G, Di Mussi R, Marangoni E, Volta CA. Can diaphragmatic ultrasonography performed during the T-tube trial predict weaning failure? The role of diaphragmatic rapid shallow breathing index. Crit Care. 2016 Sep 28;20(1):305. doi: 10.1186/s13054-016-1479-y. PMID 27677861
- [Background] Jaber S, Petrof BJ, Jung B, Chanques G, Berthet JP, Rabuel C, Bouyabrine H, Courouble P, Koechlin-Ramonatxo C, Sebbane M, Similowski T, Scheuermann V, Mebazaa A, Capdevila X, Mornet D, Mercier J, Lacampagne A, Philips A, Matecki S. Rapidly progressive diaphragmatic weakness and injury during mechanical ventilation in humans. Am J Respir Crit Care Med. 2011 Feb 1;183(3):364-71. doi: 10.1164/rccm.201004-0670OC. Epub 2010 Sep 2. PMID 20813887
- [Background] Levine S, Nguyen T, Taylor N, Friscia ME, Budak MT, Rothenberg P, Zhu J, Sachdeva R, Sonnad S, Kaiser LR, Rubinstein NA, Powers SK, Shrager JB. Rapid disuse atrophy of diaphragm fibers in mechanically ventilated humans. N Engl J Med. 2008 Mar 27;358(13):1327-35. doi: 10.1056/NEJMoa070447. PMID 18367735
- [Background] Kim WY, Suh HJ, Hong SB, Koh Y, Lim CM. Diaphragm dysfunction assessed by ultrasonography: influence on weaning from mechanical ventilation. Crit Care Med. 2011 Dec;39(12):2627-30. doi: 10.1097/CCM.0b013e3182266408. PMID 21705883
- [Derived] Demoule A, Fosse Q, Mercat A, Bergum D, Virolle S, Bureau C, Mellemseter M, Guichou R, Similowski T, Dres M, Mortaza S. Operator independent continuous ultrasound monitoring of diaphragm excursion predicts successful weaning from mechanical ventilation: a prospective observational study. Crit Care. 2024 Jul 16;28(1):245. doi: 10.1186/s13054-024-05003-0. PMID 39014512